CLINICAL TRIAL: NCT01790763
Title: Prospective,Randomized, Parallel Study to Compare the Efficacy of Mepilex and Keramatrix in Promoting Healing of Second Degree Burn Wounds
Brief Title: Compare the Efficacy of Mepilex and Keramatrix in Second Degree Burn Wounds
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to lack of funding from the sponsor this study is being withdrawn.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Keraplast Technologies, LLC (Unknown); Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-203
Record Dates: First submitted 2012-11-13; First posted 2013-02-13 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Skin Burn Degree Second
Keywords: Burn; Second-degree
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Keramatrix (Active Comparator): Keramatrix
  Interventions: Device: Keramatrix
- Mepilex (Active Comparator): Mepilex
  Interventions: Device: Mepilex

INTERVENTIONS:
Device: Keramatrix — Dressing for second degree burn
  Arms: Keramatrix
Device: Mepilex — Dressing for second degree wound
  Arms: Mepilex

SUMMARY:
The purpose of this study is to determine the extent to which Keramatrix dressing promotes the healing of second-degree burn wounds in pediatric patients.

DETAILED DESCRIPTION:
Efficacy in promoting wound healing will be determined through comparison to Mepilex, an established burn wound dressing.

ELIGIBILITY:
Inclusion Criteria:

patient age 0-18 years old Flame or scald burn 10-30% total body surface area burned Partial-thickness second-degree burns Admission within 72 hours of burn injury Clean non-infected wound as diagnosed by the attending physician

Exclusion Criteria:

* Patient older than 18
* Causes other than flame or scald injuries (ie.chemical or frostbite)
* Wounds noted to be contaminated or infected
* Patients who have received previous treatment efforts (topical dressings or previous wound debridement)
* Pregnancy lactation
* Co-morbidity which may compromise healing: known history of AIDS, ARC, HIV, cancer, autoimmune diseases,cirrhosis, tuberculosis, chronic glucocorticoid therapy, diabetes mellitus, renal insufficiency, hepatic disease, congestive heart failure prior to burn injury, associated severe head injury requiring specific treatment
* known allergy to sheep's wool

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Wound Healing | Duration of hospital stay, an expected average of 0.75 days per every percent burn until wound heals
  Wound healing will be determined by measuring wound surface area. Wound surface area will be determined through planimetry, which will be performed on digital photographs of the wounds.

SECONDARY OUTCOMES:
Infection rates | Duration of hospital stay, an expected average of 0.75 days per percent burn until wound heals
  Subjects will be monitored for unusual occurences, including signs and symptoms of infection.
Scarring | 52 weeks up to 78 weeks
  Scarring will be evaluated using the Vancouver Clinical Scar Scale. Assessments of graft pigmentation, vascularity, pliability and height will be performed at follow-up visits.
Pain | duration of hospital stay, an expected average of 0.75 days per every percent burn until wound heals, up to 3 times a week during dressing changes
  Pain will be assessed using pain scales according to age.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Jimenez, MD, Principal Investigator — University of Texas
Locations (1):
- Shriners Hospitals for Children, Galveston, Texas, United States